CLINICAL TRIAL: NCT00422565
Title: Comparison of the Efficacy and Safety of Zotarolimus-Eluting Stent Versus Sirolimus-Eluting Stent Versus PacliTaxel-Eluting Stent for Acute Myocardial Infarction Patients
Brief Title: Zotarolimus-Versus Sirolimus-Versus PacliTaxel-Eluting Stent for Acute Myocardial Infarction Patients
Acronym: ZEST-AMI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The recruitment rate was much slower than expected.
Sponsor: Seung-Jung Park (Other)
Collaborators: Cordis US Corp. (Industry); CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Professor, Cardiology, Asan Medical Center Heart Institute, Valvular Heart Disease Center, Ischemic Heart Disease Center, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006-0137
Record Dates: First submitted 2007-01-16; First posted 2007-01-17 (Estimated); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Myocardial Infarction
Keywords: Coronary Artery Disease; Stent; Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Endeavor (Experimental): Zotarolimus-eluting stent
  Interventions: Device: Endeavor, Medtronic
- Cypher (Active Comparator): Sirolimus-eluting stent
  Interventions: Device: Cypher, Cordis
- Taxus (Active Comparator): Paclitaxel-eluting stent
  Interventions: Device: Taxus Liberte, Boston Scientific

INTERVENTIONS:
Device: Endeavor, Medtronic — Zotarolimus-eluting stent
  Other Names: Zotarolimus-eluting stent
  Arms: Endeavor
Device: Cypher, Cordis — Sirolimus-eluting stent
  Other Names: Sirolimus-eluting stent
  Arms: Cypher
Device: Taxus Liberte, Boston Scientific — Paclitaxel-eluting stent
  Other Names: Paclitaxel-eluting stent
  Arms: Taxus

SUMMARY:
The trial has the following primary objective:

To compare the safety and effectiveness of primary acute MI intervention with ABT 578-eluting balloon expandable stent (Medtronic, Minneapolis, MN) vs. sirolimus-eluting balloon expandable stent (Cordis Johnson & Johnson, Warren, New Jersey) vs. paclitaxel-eluting stent (Taxus Liberte, Boston Scientific).

DETAILED DESCRIPTION:
Previous studies have documented that a slow-release polymeric sirolimus-eluting stent (Cypher, Cordis) and paclitaxel-eluting stent (Taxus, Boston Scientific) reduce neointimal formation and result in decrease of angiographic restenosis and target lesion revascularization at 1-3 years in the multicenter randomized clinical trials RAVEL, SIRIUS, and TAXUS I-VI. From these studies, the two leading drug-eluting stents (DESs) of the Cypher and Taxus have been widely and rapidly accepted as a standard treatment of coronary lesions.

Recently, randomized studies were conducted to reveal different outcomes of the different two DESs. These studies showed that the sirolimus-eluting stent was better than the paclitaxel-eluting stent in terms of lower angiographic restenosis rate or the two DESs were similar in angiographic outcomes. A recent meta-analysis supported results of the former randomized studies. Patients receiving sirolimus-eluting stent had a significantly lower risk of restenosis and target vessel revascularization compared with those receiving paclitaxel-eluting stent.

With a recent approval of new DES, ABT-578-eluting stent (Endeavor, Medtronic, Minneapolis, MN), other comparison studies have been conducted to compare Endeavor ABT-578-eluting stent with the sirolimus-eluting stent and paclitaxel-eluting stent. The ENDEAVOR clinical trials are currently in progress to evaluate a phosphoryl choline (PC)-coated ABT-578-eluting stent for the prevention of restenosis. Angiographic analysis at 4 months in the 100-patient focal de novo lesion ENDEAVOR I feasibility study demonstrated a mean in-stent percent diameter stenosis of approximately 14% and a late lumen loss of 0.3 mm with a low frequency of target lesion revascularization (1%). The clinical outcomes from the ENDEAVOR II (1,197 patients randomized to ABT-578 or bare metal stent) showed superior efficacy of the PC-coated ABT-578-eluting stent than bare-metal stent.

In patients with acute myocardial infraction (MI), routine stent implantation has been shown to have a better procedural success rate and clinical outcome than balloon angioplasty [11]. However, restenosis and vessel reocclusion remain major challenges limiting the long-term success of percutaneous treatment.

In a clinical study of 400 patients with stent implantation in acute MI, angiographic restenosis occurred in 31%, considerably more than expected for patients with stable coronary disease. There is very little information available as to the efficacy and long-term safety of DES in acute MI. The results from the several registry and randomized trials (Cypher-AMI, Typhoon, PASSION) demonstrated the short-term or long-term safety and efficacy of DES compared to BMS.

The incomplete evidence to date is that implantation of SES in patients with Acute MI is safe and effective more than BMS and results of implantation of PES are at variance with the results of the BMS. However, up to date, there are randomized trials to compare the efficacy and safety among commonly used DES (zotarolimus- vs. sirolimus- vs. paclitaxel-eluting stents) for the treatment of acute MI patients. The results of large randomized trials and larger registries will allow us to make evidence-based decisions about which stent to use in patients with acute MI. Therefore, we designed a randomized, controlled, partially blinded trial comparing the safety and efficacy of the zotarolimus vs. sirolimus vs. paclitaxel stents in acute MI patients undergoing percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be at least 18 years of age.
2. Culprit de novo lesion in a native coronary artery with significant stenosis (>50% by visual estimate) eligible for stent implantation (no limitation on stent length)
3. Prolonged, continuous (≥ 20 min) chest pain despite nitrate and: (1) at least 1mm ST-segment elevation in at least 2 leads or reciprocal ST-segment depression ≥ 2 contiguous precordial leads, or (2) newly developed left bundle branch block
4. Symptoms < 12 hours
5. The patient or guardian agrees to the study protocol and the schedule of clinical and angiographic follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

1. The patient has a known hypersensitivity or contraindication to any of the following medications:

   * Heparin
   * Aspirin
   * Both Clopidogrel and TIclopidine
   * Sirolimus, paclitaxel, ABT 578
   * Stainless steel and/or
   * Contrast media (patients with documented sensitivity to contrast which can be effectively pre-medicated with steroids and diphenhydramine [e.g. rash] may be enrolled. Patients with true anaphylaxis to prior contrast media, however, should not be enrolled).
2. Systemic (intravenous) Sirolimus, paclitaxel or ABT-578 use within 12 months.
3. Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study.
4. History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or will refuse blood transfusions.
5. Fibrinolytic therapy for current MI treatment
6. Previous coronary intervention on target vessel
7. Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
8. Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
9. Previously documented LVEF <30%.
10. Evident cardiogenic shock before randomization
11. Patients with left main stem stenosis (>50% by visual estimate)
12. Severe calcification or tortuosity
13. Multi-vessel disease with non-culprit vessel requiring bypass surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2006-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The composite of death (all cause-mortality), MI (Q wave and non Q wave) and ischemia-driven target vessel revascularization. | At 12 months after the index procedure

SECONDARY OUTCOMES:
All-cause Death | 1 month, 6 month, 1 year and thereafter annaully up to 5 years
Cardiac death | 1 month, 6 month, 1 year and thereafter annaully up to 5 years
Recurrent Myocardial infarction | 1 month, 6 month, 1 year and thereafter annaully up to 5 years
Target vessel revascularization (all and ischemia-driven) | 1 month, 6 month, 1 year and thereafter annaully up to 5 years
Target lesion revascularization (all and ischemia-driven) | 1 month, 6 month, 1 year and thereafter annaully up to 5 years
Stent thrombosis for the patients | 1 month, 6 month, 1 year and thereafter annaully up to 5 years
Late luminal loss in both in-stent and in-segment | at 8 month angiographic follow-up
Binary restenosis in both in-stent and in-segment | at 8 month angiographic follow-up
Procedural success defined as achievement of a final diameter stenosis of <30% by QCA using any percutaneous method, without the occurrence of death, Q wave MI, or repeat revascularization of the target lesion | during the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Department of Medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (12):
- South Korea (12):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Daegu Catholic University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Asan Medical Center, Gangneung
  - Chonnam National University Hospital, Gwangju
  - NHIC Ilsan Hospital, Ilsan
  - Pusan Natioanal University Hospital, Pusan
  - Asan Medical Center, Seoul
  - Korea University Hospital, Seoul
  - St. Mary's Catholic Medical Center, Seoul
  - Ulsan University Hospital, Ulsan
  - Yonsei University Wonju Christian Hospital, Wŏnju